CLINICAL TRIAL: NCT04750434
Title: PET MRI as a Staging Tool for Head and Neck Cancer
Status: Completed | Type: Observational
Sponsor: Hoag Memorial Hospital Presbyterian (Other)
Responsible Party: Sponsor
Other Study IDs: 161-19-HC
Record Dates: First submitted 2021-02-08; First posted 2021-02-11 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Head Cancer; Neck Cancer
Keywords: head cancer; neck cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To explore the use of PET/MRI in the staging and pretreatment evaluation of patients with head and neck cancer and to compare this modality to standard PET/CT imaging.

DETAILED DESCRIPTION:
This study is a prospective clinical study whereby an emerging technology, PET/MRI will be compared to a more standard imaging modality, PET/CT, using newly diagnosed head and neck cancer patients as subjects. PET/MRI will also be used in this study to explore the merits of this new technology in determining extent of disease, functional impact, and potential treatment outcome.

In this study, subjects suitable for enrollment will be identified by the investigators involved in the study. These subjects will be identified through contact with these investigators and referred for enrollment per protocol. This protocol will include determining enrollment suitability based on inclusion and exclusion criteria. Once accepted as a candidate for the study, the newly diagnosed head and neck cancer patients will undergo both PET/CT and PET/MRI imaging within one week of each other. These studies will then be reviewed by a radiologist specializing in Head and Neck radiology familiar with PET imaging. The studies will be compared for any imaging differences. The imaging findings will then be correlated with pathological findings after surgery to determine if there are any consistent findings that correlate with adverse pathological findings, if found.

The specific imaging data points to be determined by a radiologist will be tumor and metastatic disease size, SUV uptake, specific anatomic structures involved with tumor, imaging irregularities and characteristics of those imaging irregularities of the involved structures locally and regionally (if present), imaging characteristics of the different phases of MRI (T1, T2, etc.), and any other notable imaging characteristic.

ELIGIBILITY:
Inclusion Criteria:

* Active head and neck cancer that require PET/CT regardless of the point of treatment
* TNM staging I or II

Exclusion Criteria:

* Patients whose primary treatment option is chemotherapy or radiation therapy (not surgical)
* Implanted pacemakers
* Intracranial aneurysm clips
* Cochlear implants
* Certain prosthetic devices
* Implanted drug infusion pumps
* Neurostimulators
* Bone-growth stimulators
* Certain intrauterine contraceptive devices; or
* Any other type of iron-based metal implants.
* MRI should not also be used on persons with the presence of internal metallic objects such as bullets or shrapnel, as well as surgical clips, pins, plates, screws, metal sutures, or wire mesh.
* Subject with breast tissue expanders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who are referred to Hoag for imaging services related to Head and Neck cancer will be recruited.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2020-03-03 (Actual); Primary Completion 2024-08-16 (Actual); Study Completion 2024-08-16 (Actual)

PRIMARY OUTCOMES:
PET MRI as a Staging Tool for Head and Neck Cancer | 18 months
  Outcomes from this study will include a comparison of PET/MRI with PET/CT directly in a series of patients where surgical pathology specimens are available for correlation.

CONTACTS AND LOCATIONS:
Locations (1):
- Hoag Memorial Hospital Presbyterian, Newport Beach, California, United States